CLINICAL TRIAL: NCT04189003
Title: Identification of Specific Molecular Signatures by Capture-HPV and Next-generation Sequencing in HPV-induced Oropharyngeal Cancers
Brief Title: Molecular Signatures of HPV+ ORL Cancers (OROPAP)
Acronym: OROPAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180166; APHP180166 (Other: AP-HP)
Record Dates: First submitted 2019-10-18; First posted 2019-12-06 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Oropharyngeal Cancer; Human Papillomavirus-Related Carcinoma
Keywords: ORL Cancers; HPV+ tumor; molecular signature; human papillomavirus
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Frozen and/or FFPE biopsies of HPV-positive oropharyngeal tumors and frozen blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify HPV molecular signature in head and neck cancer to establish a new classification for positive human papillomavirus oropharyngeal tumor

DETAILED DESCRIPTION:
OROPAP is a monocentric exploratory study with retrospective inclusion of patients.

The retrospective study focus on patients who have had surgery for HPV-positive oropharyngeal tumors whose survival is at least 2 year.

Frozen and or FFPE biopsies of these tumors and frozen blood samples are available via the HEGP biological resources platform.

The HPV molecular signatures will be identified by the capture-HPV technique.

For each patient, clinical-anatomo-pathological data such as tumor size, tumor stage, presence or absence of metastasis, histological stage, different treatment lines and 2-years survival data will be collected through the use of data warehouse available on the HEGP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HPV + oropharyngeal cancer

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV-induced oropharyngeal cancer with survival follow-up greater than 2 years
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Description the HPV molecular signatures identified by the Capture-HPV technique and comparison of these signatures with those already described in the classification described in the Holmes et al. in the cervix | 18 months
  Establish a new classification based on HPV molecular signature for positive human papillomavirus oropharyngeal tumor

SECONDARY OUTCOMES:
Quantification of HPV circulating tumoral DNA in peripheral blood by droplet based digital PCR | 18 months
  Find in the peripheral blood of patients, the presence of circulating tumoral HPV DNA (ctDNA) by droplet based digital PCR and when it is possible compare chromosomal insertion patterns of HPV ct DNA as those found in tumors
Correlate identified HPV molecular signature with clinical-anatomo-pathological data. | 18 months
  Look for an association between the presence of specific HPV molecular signatures and clinical-anatomo-pathological data.
Number of Death of any cause, or eventual relapse | 18 months
  Look for an association between the presence of these molecular signatures and the survival of patients.
Ratio of the number of copies of viral genes to the number of cells | 18 months
  Measure the viral load of HPV in the tumor.
Precise description of HPV insertion localisation in human genome when HPV is integrated | 18 months
  Identify disrupted metabolic pathways in tumor cells.
Description of new HPV viral variants based on complete HPV genome sequencec obtained by Capture-HPV coupled with NGS | 18 months
  Analyze of complete viral genomes and identify potential variants through sequencing data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hélène PÉRÉ, PhD, Study Director — AP-HP, Hôpital Européen Georges Pompidou
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in publication could be shared. Individual participant data detailed in meta analysis protocol could be shared
Supporting Information: Study Protocol, ICF
Time Frame: one year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization